CLINICAL TRIAL: NCT01899170
Title: Towards Individualized Deep Brain Stimulation Treatment of Chronic Neuropathic Pain
Acronym: DBSforPain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Device for multi coil TMS no longer supported
Sponsor: University of Aarhus (Other)
Collaborators: Stanford University (Other); California Pacific Medical Center Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 28052013; 2013-002385-39 (EudraCT Number)
Record Dates: First submitted 2013-07-03; First posted 2013-07-15 (Estimated); Last update posted 2021-09-14 (Actual); Status verified 2013-07

CONDITIONS: Neuralgia
Keywords: deep brain stimulation; multi-coil transcranial magnetic stimulation; PET-imaging; personalized treatment
MeSH Terms: conditions — Neuralgia | interventions — Deep Brain Stimulation; carfentanil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sham-DBS (Sham Comparator): Only patients. Inactive deep brain stimulation for the initial three months following implantation.
  Interventions: Procedure: Deep brain stimulation; Device: Cervel Neurotech, Multi-coil TMS; Drug: 11C-Carfentanil
- Active DBS (Active Comparator): Only patients. Active deep brain stimulation for the initial three months following surgery.
  Interventions: Procedure: Deep brain stimulation; Device: Cervel Neurotech, Multi-coil TMS; Drug: 11C-Carfentanil
- TMS and PET imaging (Experimental): This experiment includes all participants (cases and controls). Each subject will undergo both active and sham stimulation (cross-over) with Cervel Neurotech Multi-coil TMS and related test/re-test PET imaging with 11C-Carfentanil. Only patients will proceed into deep brain stimulation experiments.
  Interventions: Device: Cervel Neurotech, Multi-coil TMS; Drug: 11C-Carfentanil

INTERVENTIONS:
Procedure: Deep brain stimulation — Implantation of a deep brain stimulation electrode into pain processing brain areas
  Arms: Active DBS; Sham-DBS
Device: Cervel Neurotech, Multi-coil TMS — Non-invasive selective stimulation of deep brain areas using magnetic fields.
  Other Names: TMS
Drug: 11C-Carfentanil — PET-radioligand for functional brain imaging to assess opioid binding. The compound is a potent synthetic opioid.
  Other Names: 11C-Carfentanyl

SUMMARY:
Chronic neuropathic pain affects millions of individuals worldwide. It causes marked reduction of health, utility and quality of life and represents a considerable economic burden to society due to loss of work capacity and large treatment expenses. The proposed project will explore new and rational methods for deep brain stimulation treatment of patients with severe chronic neuropathic pain, resistant to conventional treatment. Deep brain stimulation is a neurosurgical procedure in which a small stimulating electrode is implanted into deep brain areas. Furthermore, we will utilize new positron emission tomography neuroimaging and a new prototyped technology, called targeted transcranial magnetic stimulation, to predict the outcome of deep brain stimulation and localize brain regions with maximum symptom relief for each patient. This will optimize the selection of patients for deep brain stimulation and provide a rational customized choice of brain target for each patient, without surgical intervention. Novel techniques will be validated on healthy volunteers and at the same time provide new insights into the mechanisms underlying brain stimulation and pain perception. The project has great clinical impact, potential for innovative development and industrial spin-out, facilitates exchange for Danish research talents and senior researchers with Stanford University and California Pacific Medical Research Institute in San Francisco, and unites world leading experts in pain research and clinical treatment to achieve its goals.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria (case and control):

* No gender criteria
* Age > 25 years.
* Legal competency.
* Ability to comply with the proposed protocol schedule.
* Stability of chronic medical diseases.
* A negative validated pregnancy test for fertile female participants prior to project enrolment.
* Use of validated anti-conception for fertile female participants

Case-specific inclusion criteria:

* Well-defined neuropathic pain [21].
* Chronic and stable pain condition. Numerical Rating Scale score > 5.
* Documented resistance to, or poor tolerance of pharmacological treatments. Unless contraindicated, the treatment must have included opiate derivatives, tri-cyclic antidepressants and anti-epileptic drugs.

Exclusion Criteria:

General exclusion criteria:

* Pregnancy or nursing.
* Cognitive impairment.
* Alcohol or drug abuse
* Severe psychiatric disorders.
* Allergies towards compounds used in the trial, such as PET tracers, Capsaicin, etc. Other significant medical allergies.
* Severe medical disorders
* Neurodegenerative disorders
* Severe cerebrovascular diseases and risk-factors, malignant hypertension, vascular abnormalities.
* Prior intracranial surgery
* Cardiac pacemaker or other implanted electronic medical devices
* Coagulopathy (excl. drug induced)
* Structural brain abnormalities
* Epilepsy or prior isolated seizure.
* Severe obesity
* Severe claustrophobia
* Magnetic metallic implants
* Other conditions that may contraindicate deep brain stimulation surgery, full anesthesia, transcranial magnetic stimulation, PET/CT imaging (specifically the use of carfentanil) or magnetic resonance imaging. This will be evaluated according to specific investigational product specifications and clinical guidelines.

Control specific exclusion criteria:

- Chronic pain syndrome

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Pain relief upon deep brain stimulation of the dorsal anterior cingulate cortex. | Assessment after 3 and 12 months of active stimulation
  We will measure the changes in pain ratings upon deep brain stimulation of the dorsal anterior cingulate gyrus. Results will be based on the numerical rating scale and validated questionnaires. We will compare active and sham stimulation and changes upon activation of initial sham-stimulation.
Predictive values of PET imaging and transcranial magnetic stimulation on deep brain stimulation outcome | Assessed upon final evaluation of deep brain stimulation outcome (expected 2 years)
  Individuals will be classified according to PET activity/no-activity and positive/null-negative outcome of transcranial magnetic stimulation. We will correlate the effect of deep brian stimulation to these categories and evaluate their predictive values.

SECONDARY OUTCOMES:
Effect of deep brain stimulation on cingulate opioid binding and blood flow. | After 3 and 12 months of active deep brain stimulation
  We will do test/re-test PET imaging before and after deep brain stimulation surgery to assess the effect of this treatment on cingulate opioid binding and blood flow. We will utilize 11C-Carfentanil and 15O-water PET, respectively.
Pain relief upon individualized deep brain stimulation | After 3 and 12 months of active deep brain stimulation
  Patients that derive no benefit from initial deep brain stimulation treatment of the dorsal anterior cingulate, will be offered deep brain stimulation of another expectedly efficacious brain area. The choice of target will be based of PET images and magnetic stimulation testing. Results of deep brain stimulation will be based on the numerical rating scale and validated pain questionnaires.

OTHER OUTCOMES:
Effect of transcranial magnetic stimulation on pain ratings, cingulate opioid binding and blood flow | results will be assessed upon final transcranial magnetic stimulation session (last participant/last treatment, average 5 weeks)
  We will do test/re-test PET imaging with transcranial magnetic stimulation in between. We will evaluate quantitative effects on 1) pain ratings using the numerical rating scale, 2) cingulate opioid binding using 11C-carfentanil PET and 3) cingulate blood flow using 15O-water PET. Results will be compared for sham stimulation and active stimulation in each individual, and also between cases and controls.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Christian H Sørensen, MD,PhD,DMSc, Principal Investigator — Aarhus University Hospital, Department of Neurosurgery
Locations (1):
- Aarhus University Hospital, Aarhus, Central Jutland, Denmark